CLINICAL TRIAL: NCT04698785
Title: A Multicentre Phase II Study of Efficacy of Regorafenib as Maintenance Treatment in Patients With High Grade Bone Sarcomas at Diagnosis or Relapse and Without Complete Remission After Standard Treatment
Brief Title: Efficacy of Regorafenib Combined With Best Supportive Care as Maintenance Treatment in High Grade Bone Sarcomas Patients
Acronym: REGOMAIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET19000144 (REGOMAIN)
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Bone Sarcoma; Osteosarcoma
Keywords: Bone sarcoma; Osteosarcoma; Maintenance therapy; Regorafenib; Progression-free rate; Objective response rate; Disease control rate; Overall survival; Quality of life; Tolerance; Tyrosine inhibitor kinase; Multitarget inhibitor; High-grade; Progression-Free survival
MeSH Terms: conditions — Bone Neoplasms; Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib and best supportive care (Experimental): Treatment will be divided in 28 days cycles, including a 21-day period of treatment by regorafenib and best supportive care followed by a 7-day period of rest.
  In case of toxicity, dose can be reduced or treatment interrupted according to Specific Product Characteristics (SPC).
  Patients can receive up to a maximum of 13 cycles (maximum treatment period : 12 Months).
  Interventions: Drug: Treatment by regorafenib and best supportive care

INTERVENTIONS:
Drug: Treatment by regorafenib and best supportive care — Treatment for 13 cycles (12 months) maximum.
  During each cycle :
  * patients ≥ 16 years old and patients <16 old with Body Surface Area (BSA) ≥ 1,70 m2 will take 3 tablets, once a day, corresponding to a total of 120 mg Regorafenib, during 21 days, followed by 7 days without treatment.
  * patients < 16 years old with a 1,30 m2 ≤ BSA ≥ 1,70 m2 will take 2 tablets, once a day, corresponding to a total of 80 mg Regorafenib, during 21 days, followed by 7 days without treatment
  Other Names: Experimental arm

SUMMARY:
This is a multicenter phase II study concerning patients with high-grade bone sarcoma (HGBS) without complete remission after standard treatment at diagnosis or at relapse.

Patients will be treated with regorafenib + best supportive care (BSC) for a maximum of 12 months as maintenance therapy after standard line therapy completion.

Progression free rate (PFR) data will be collected and analysed for all included patients to evaluate if regorafenib + BSC can be considered as an interesting treatment for further investigations in this indication.

DETAILED DESCRIPTION:
This is a multicenter phase II study.

Patients with evaluable unresectable residual disease will be accrued after they completed standard of care, consisting of:

* At diagnosis: standard multimodal treatment based on histological subtype
* At relapse: chemotherapy

Patients who meet the eligibility criteria will receive regorafenib + best supportive care (BSC) as maintenance treatment for a maximum 12 months period.

After their eligibility has been confirmed, patients will receive regorafenib until disease progression, or for a maximum of 12 months, or unacceptable toxicity or willingness to stop, whichever occurs first.

After the completion of the maintenance therapy (12 months) patients will be followed-up until the first radiological disease progression, unless a premature disease progression occurred. All patients will be followed-up until the data cut-off (12 months after the last inclusion).

The vital status will be updated once for all patients at 24 months after the last inclusion, based on patient's medical file.

ELIGIBILITY:
INCLUSION CRITERIA:

I1. Age ≥ 12 years at the day of consenting to the study;

I2. Patients must have histologically confirmed high-grade sarcomas of bone primary localisation, including but not limited to: Osteosarcomas, Ewing sarcomas, Chondrosarcomas, Undifferenciated Pleomorphic Sarcomas (UPS), Leiomyosarcomas (LMS) and Angiosarcomas

I3. Evaluable residual disease not amenable to resection after multimodal treatment principles either at diagnosis (after standard multimodal treatment based on the histological subtype) or at relapse (chemotherapy)

I4. Non progressive disease (defined by the investigator according to the RECIST version 1.1 Appendix 1) at study entry;

I5. Interval between the date of last anticancer treatment (chemotherapy or surgery) and the start date of regorafenib: at least 4 weeks but no longer than 2 months;

I6. Life expectancy of greater than 6 months;

I7. Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky ≥ 70%) (Appendix 2);

I8. Adequate bone marrow and organ function defined by the following laboratory results:

a. Bone marrow: i. Absolute neutrophil count ≥ 1.5 Giga/l ii. Platelets ≥ 100 Giga/l iii. Haemoglobin≥ 9 g/dl

b. Hepatic function: i. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x Upper Limit of Normal (ULN) (≤ 5.0 × ULN for patients with liver involvement of their cancer) ii. Bilirubin ≤1.5 X ULN iii. Alkaline phosphatase ≤ 2.5 x ULN (≤ 5 x ULN in patient with liver involvement of their cancer). If Alkaline phosphatase > 2.5 ULN, hepatic isoenzymes 5-nucleotidase or gamma-glutamyltransferase (GGT) tests must be performed; hepatic isoenzymes 5-nucleotidase must be within the normal range and/or GGT < 1.5 x ULN.

c. Renal function: i. Serum creatinine ≤ 1.5 x ULN ii. Glomerular Filtration Rate (GFR) ≥ 30 ml/min/1.73m2 according to the Modified Diet in Renal Disease (MDRD) abbreviated formula iii. Spot urine must not show ≥ 1 "+" protein in urine or the patient will require a repeat urine analysis. If repeat urinalysis shows 1 "+" protein or more, a 24-hour urine collection will be required and must show total protein excretion < 1000 mg/24 hours

d. Coagulation: International Normalized Ratio (INR)/Partial Thromboplastin Time (PTT) ≤1.5 x ULN; Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care;

e. Pancreatic function: Lipase ≤ 1.5 x ULN

I9. Recovery to anticancer-treatment related NCI-CTCAE v5 Grade 0 or 1 level or recovery to baseline preceding the prior treatment from any previous drug/procedure related toxicity (except alopecia, anaemia, and hypothyroidism);

I10. Women of childbearing potential and male patients must agree to use adequate contraception (including at least the use of condoms) for the duration of treatment and for 7 months (210 days) in women of childbearing potential or 4 months (120 days) in men sexually active with women of childbearing potential after the last dose of regorafenib

I11. Patients, and their parents when applicable, must sign and date an informed consent document indicating that they have been informed of all the pertinent aspects of the trial prior to enrolment;

I12. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures;

I13. Patients affiliated to the Social Security System

I14. Body Surface Area (BSA) ≥ 1.30m² at the time of consenting to the study

EXCLUSION CRITERIA:

E1. Prior treatment with any VEGFR inhibitor (thus, any prior exposure to regorafenib, sunitinib, sorafenib, pazopanib, bevacizumab, or other VEGFR inhibitor);

E2. All soft tissue sarcomas (including but not limited to soft tissue osteosarcoma), and chordomas;

E3. Prior history of malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) within 3 years prior to randomization;

E4. Cardiovascular dysfunction defined by:

* Left ventricular ejection fraction (LVEF) < 50%,
* Congestive heart failure ≥ New York Heart Association (NYHA) class 2,
* Myocardial infarction < 6 months prior to first study drug administration,
* Cardiac arrhythmias requiring therapy (beta blockers or digoxin are permitted),
* Unstable (angina symptoms at rest) or new-onset angina within the last 3 months prior to first study drug administration;
* Uncontrolled hypertension (systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg despite optimal treatment);
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the last 6 months before the first study drug administration;

E5. Major surgical procedure, open biopsy or significant traumatic injury within 28 days before the first study drug administration;

E6. Ongoing infection > Grade 2 according to NCI-CTCAE v5;

E7. Known history of human immunodeficiency virus infection;

Nota Bene: Subjects with diagnosed human immunodeficiency virus (HIV) are eligible to participate in the study if they meet the following criteria :

1. No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months prior to enrolment;
2. No history of AIDS-defining cancers (e.g. Kaposi's sarcoma, aggressive B-cell lymphoma and invasive cervical cancer);
3. Subjects should be on established anti-retroviral therapy for at least 4 weeks and have an HIV viral load of < 400 copies/mL prior to enrolment;

E8. Active or chronic hepatitis B or C requiring treatment with antiviral therapy; Nota Bene: Subjects with a history of hepatitis B or C who have normal alanine aminotransferase (ALT) and are hepatitis B surface antigen negative and/or have undetectable HCV RNA are eligible

E9. Dehydration according to NCI-CTCAE v5 Grade >1;

E10. Difficulties to swallow oral medication and/or any mal-absorption condition and/or any Gastrointestinal (GI) disease that may significantly alter the absorption of regorafenib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small bowel resection);

E11. Patients with seizure disorder requiring medication;

E12. Concurrent enrolment in another clinical trial in which investigational therapies are administered;

E13. Known hypersensitivity to the active substance or to any of the excipients;

E14. Pregnant women, women who are likely to become pregnant or are breast-feeding. Women of childbearing potential must have a negative serum β-Human Chorionic Gonadotropin (HCG) pregnancy test within 7 days prior randomization;

E15. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;

E16. Patients with history of non-compliance to medical regimens or unwilling or unable to comply with the protocol;

E17. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent;

E18. Non-healing wound, non-healing ulcer, or non-healing bone fracture;

E19. Patients with evidence or history of any bleeding diathesis, irrespective of severity;

E20. Any haemorrhage or bleeding event ≥ CTCAE v5 Grade 3 within 4 weeks prior to the first study drug administration;

E21. Clinically significant unrelated systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results;

E22. Patients using prohibited concomitant and/or concurrent medications (see section "Prohibited concomitant/concurrent treatments);

E23. Patients under tutorship or curatorship.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Rate at 4 months (4m-PFR) | Up to 16 weeks after the date of regorafenib + BSC treatment initiation
  The Progression-Free Rate at 4 months (4m-PFR) will be defined as the proportion of patients with a complete response, a partial response or stable disease, confirmed on tumour assessments according to the RECIST V1.1 at 4 months (16 weeks) after the date of regorafenib + BSC treatment initiation.
  Patients with a non-progressive disease at 16 ± 2 weeks after the date of regorafenib + BSC treatment initiation will be considered as "success" patients.
  Patients with a progressive disease and patients who died from any cause at 16 ± 2 weeks after the date of regorafenib + BSC treatment initiation will be considered as "failure" patients.
  At the time of analysis, if at least 18 "successes" are observed among the 36 analyzed patients, the regorafenib + BSC treatment will be considered as interesting for further investigations in this indication.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years
  PFS will be described from date of regorafenib + BSC treatment initiation to the date first documented disease progression according to RECIST V1.1 or the date of death due to any cause.
  Patients alive without progression at the time of data cut-off will be censored at the time of latest tumour evaluation.
Objective Response Rate (ORR) | Up to 3 years
  The Objective Response Rate (ORR) will be defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) (RECIST V1.1)
Disease Control Rate (DCR) at 2 months | 2 months
  The Disease Control Rate (DCR) will be defined as the proportion of patients with a best overall response of CR, PR or Stable Disease (SD) (RECIST V1.1) 2 months after randomization
Disease Control Rate (DCR) at 4 months | 4 months
  The Disease Control Rate (DCR) will be defined as the proportion of patients with a best overall response of CR, PR or Stable Disease (SD) (RECIST V1.1) 4 months after randomization
Overall Survival (OS) | Up to 3 years
  The Overall Survival (OS) will be defined as the time from date of regorafenib +BSC treatment initiation to the date of death, from any cause. Patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Quality of Life (QoL) | Up to 1 year
  The patient's Quality of Life (QoL) will be assessed using the EORTC Quality Of Life Questionnaire (QLQ)-C30 file. Scores will be calculated at each time point according to the scoring manuals. Descriptive statistics will be used to evaluate baseline scores and evolution of scores from baseline to each time point. Data will be compared between arms using the Student's t-test. The QoL data will also be presented graphically if deemed relevant.
Tolerance profile of treatment | Up to 3 years
  The safety will be described mainly on the frequency of adverse events (AE) coded using the common toxicity criteria (NCI-CTCAE v5.0) grade. Descriptive statistics will be provided for characterizing and assessing patient tolerance to treatment. AE will be coded according to the MedDRA®.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi BRAHMI, Principal Investigator — Centre Léon Bérard, Lyon
Locations (16):
- France (16):
  - Chu Besancon, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de La Timone, Marseille
  - Icm Val D'Aurelle, Montpellier
  - Hotel Dieu Nantes, Nantes
  - Institut Curie, Paris
  - Hôpital COCHIN, Paris
  - Ico Rene Gauducheau, Saint-Herblain
  - Chu Saint-Etienne, Saint-Priest-en-Jarez
  - CHRU Hôpital Hautepierre, Strasbourg
  - ICANS, Strasbourg
  - Iuct Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif